CLINICAL TRIAL: NCT00051922
Title: Evaluation of the Safety of a Polyvalent Vaccinia Virus HIV-1 Envelope Recombinant Vaccine (PolyEnv1) in Healthy Adults
Brief Title: Development of a New HIV Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Patricia Flynn, MD, St. Jude's Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P01AI045142 (NIH); P01AI045142 (NIH)
Record Dates: First submitted 2003-01-17; First posted 2003-01-22 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: HIV Infections
Keywords: HIV Preventive Vaccine; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

ARMS (1):
- 1 (Experimental): Participants will receive vaccine and will be followed for 1 year
  Interventions: Biological: PolyEnv1

INTERVENTIONS:
Biological: PolyEnv1 — Recombinant vaccinia virus vaccine

SUMMARY:
The purpose of the study is to determine the safety of a new HIV vaccine and to evaluate the immune response to the vaccine. Only some HIV genes are used to make the vaccine and therefore the vaccine cannot itself cause HIV or AIDS.

DETAILED DESCRIPTION:
HIV-1 presents several challenges to vaccine design, including: 1) high mutation rates resulting in tremendous diversity of virus envelope, the target of neutralizing antibody, such that antibody elicited to one envelope may not protect from virus with a distinct envelope; 2) envelope from infected persons differs from envelopes obtained from T-cell line cultures, the usual source of envelope for vaccines; and 3) envelope glycoprotein exists as oligomers on the virion surface, not as the monomers used in previous vaccines. This study will test a new vaccine that has been designed to meet these challenges by delivering diverse, patient-derived, oligomeric envelopes to induce multiple type-specific responses capable of recognizing native envelope on natural variants. The vaccine vector used in this vaccine trial is recombinant vaccinia virus based on the NYCDH vaccinia isolate.

Participants in this study will receive the PolyEnv1 HIV vaccine and will be followed for one year. Laboratory tests will be performed at 10 study visits to monitor the participants' immunologic response and assess the safety of the vaccine. Patients will also have numerous HIV tests throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 negative
* Availability for one year of follow-up
* No evidence of previous smallpox vaccination
* Acceptable methods of contraception

Exclusion Criteria:

* Immunosuppressive or chronic illness
* Medical or psychological conditions which could affect compliance
* High risk for HIV infection
* Live attenuated vaccines within 60 days
* Experimental agents within 30 days
* Blood products within past 6 months
* Eczema
* Pregnant or lactating women
* Household contact with immunodeficient person, pregnant woman, or child less than 12 months of age
* Allergy to gentamicin

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 1997-10; Primary Completion 2006-07 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Tolerability and safety of the PolyEnv1 vaccine | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Flynn, MD, Principal Investigator — Associate Member; Julia L. Hurwitz, PhD, Principal Investigator — Member
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Background] Brown SA, Stambas J, Zhan X, Slobod KS, Coleclough C, Zirkel A, Surman S, White SW, Doherty PC, Hurwitz JL. Clustering of Th cell epitopes on exposed regions of HIV envelope despite defects in antibody activity. J Immunol. 2003 Oct 15;171(8):4140-8. doi: 10.4049/jimmunol.171.8.4140. PMID 14530336
- [Background] Caver TE, Lockey TD, Srinivas RV, Webster RG, Hurwitz JL. A novel vaccine regimen utilizing DNA, vaccinia virus and protein immunizations for HIV-1 envelope presentation. Vaccine. 1999 Mar 17;17(11-12):1567-72. doi: 10.1016/s0264-410x(98)00355-7. PMID 10195794
- [Background] Lockey TD, Slobod KS, Caver TE, D'Costa S, Owens RJ, McClure HM, Compans RW, Hurwitz JL. Multi-envelope HIV vaccine safety and immunogenicity in small animals and chimpanzees. Immunol Res. 2000;21(1):7-21. doi: 10.1385/IR:21:1:7. PMID 10803879
- [Background] Rencher SD, Lockey TD, Srinivas RV, Owens RJ, Hurwitz JL. Eliciting HIV-1 envelope-specific antibodies with mixed vaccinia virus recombinants. Vaccine. 1997 Feb;15(3):265-72. doi: 10.1016/s0264-410x(96)00185-5. PMID 9139484
- [Background] Rencher SD, Slobod KS, Dawson DH, Lockey TD, Hurwitz JL. Does the key to a successful HIV type 1 vaccine lie among the envelope sequences of infected individuals? AIDS Res Hum Retroviruses. 1995 Sep;11(9):1131-3. doi: 10.1089/aid.1995.11.1131. No abstract available. PMID 8554911
- [Background] Richmond JF, Mustafa F, Lu S, Santoro JC, Weng J, O'Connell M, Fenyo EM, Hurwitz JL, Montefiori DC, Robinson HL. Screening of HIV-1 Env glycoproteins for the ability to raise neutralizing antibody using DNA immunization and recombinant vaccinia virus boosting. Virology. 1997 Apr 14;230(2):265-74. doi: 10.1006/viro.1997.8478. PMID 9143282
- [Background] Slobod KS, Bonsignori M, Brown SA, Zhan X, Stambas J, Hurwitz JL. HIV vaccines: brief review and discussion of future directions. Expert Rev Vaccines. 2005 Jun;4(3):305-13. doi: 10.1586/14760584.4.3.305. PMID 16026246
- [Background] Slobod KS, Coleclough C, Brown SA, Stambas J, Zhan X, Surman S, Jones BG, Zirkel A, Freiden PJ, Brown B, Sealy R, Bonsignori M, Hurwitz JL. Clade, Country and Region-specific HIV-1 Vaccines: Are they necessary? AIDS Res Ther. 2005 Apr 28;2(1):3. doi: 10.1186/1742-6405-2-3. PMID 15860130
- [Background] Surman S, Lockey TD, Slobod KS, Jones B, Riberdy JM, White SW, Doherty PC, Hurwitz JL. Localization of CD4+ T cell epitope hotspots to exposed strands of HIV envelope glycoprotein suggests structural influences on antigen processing. Proc Natl Acad Sci U S A. 2001 Apr 10;98(8):4587-92. doi: 10.1073/pnas.071063898. Epub 2001 Apr 3. PMID 11287644
- [Background] Zhan X, Slobod KS, Surman S, Brown SA, Lockey TD, Coleclough C, Doherty PC, Hurwitz JL. Limited breadth of a T-helper cell response to a human immunodeficiency virus envelope protein. J Virol. 2003 Apr;77(7):4231-6. doi: 10.1128/jvi.77.7.4231-4236.2003. PMID 12634380
- [Result] Slobod KS, Lockey TD, Howlett N, Srinivas RV, Rencher SD, Freiden PJ, Doherty PC, Hurwitz JL. Subcutaneous administration of a recombinant vaccinia virus vaccine expressing multiple envelopes of HIV-1. Eur J Clin Microbiol Infect Dis. 2004 Feb;23(2):106-10. doi: 10.1007/s10096-003-1075-3. Epub 2004 Jan 20. PMID 14735404
- See also: Click here for more information about St. Jude Children's Research Hospital. — http://www.stjude.org